CLINICAL TRIAL: NCT00313300
Title: A Phase 2, Placebo-Controlled, Randomized, Double Blind, Parallel Arm, Dose Ranging Study to Evaluate Safety and Efficacy of Apixaban in Patients With a Recent Acute Coronary Syndrome.
Brief Title: Safety Study of Apixaban in Recent Acute Coronary Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CV185-023
Record Dates: First submitted 2006-04-10; First posted 2006-04-12 (Estimated); Results first posted 2015-10-15 (Estimated); Last update posted 2015-12-30 (Estimated); Status verified 2015-11

CONDITIONS: Acute Coronary Syndrome (ACS)
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — apixaban

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- A1 (Active Comparator)
  Interventions: Drug: Apixaban
- A2 (Experimental)
  Interventions: Drug: Apixaban
- A3 (Placebo Comparator)
  Interventions: Drug: Placebo
- A4 (Experimental)
  Interventions: Drug: Apixaban

INTERVENTIONS:
Drug: Apixaban — Tablets, Oral, 2.5 mg, twice daily, 26 weeks
  Arms: A1
Drug: Apixaban — Tablets, Oral, 10 mg, once daily, 26 weeks
  Arms: A2
Drug: Placebo — Tablets, Oral, 0, twice daily, 26 weeks
  Arms: A3
Drug: Apixaban — Tablets, Oral 10 mg, twice daily, 26 weeks
  Arms: A4

SUMMARY:
The purpose of this clinical research study is to determine whether apixaban will be safe in people who have recently had unstable angina or a heart attack.

ELIGIBILITY:
Key Inclusion Criteria:

* Recent (< = 7 days) Acute Coronary Syndrome (ACS).
* Clinically stable on optimal treatment

Key Exclusion Criteria:

* High bleeding risk.
* Ongoing anticoagulant use.
* Need for chronic (>3 months) daily nonsteroidal anti-inflammatory drug (NSAID) or chronic high dose acetylsalicylic acid (ASA) use (>325 mg/day

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1741 (Actual)
Dates: Start 2006-05; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (127):
- United States (30):
  - Scottsdale Cardiovasular Research Institute, Scottsdale, Arizona
  - Los Angeles County & University Of Southern Ca. Medical Cen., Los Angeles, California
  - Radiant Research,Santa Rosa, Santa Rosa, California
  - South Denver Cardiology Associates, Littleton, Colorado
  - Watson Clinic Center For Research, Lakeland, Florida
  - Heart & Vasc Inst Of Fl, Safety Harbor, Florida
  - Indian River Medical Center, Vero Beach, Florida
  - Cardiac Disease Specialists, P.C., Atlanta, Georgia
  - Georgia Heart Specialists, Covington, Georgia
  - Heartcare Midwest, Peoria, Illinois
  - The Care Group, Llc., Indianapolis, Indiana
  - Iowa Heart Center, Des Moines, Iowa
  - University Of Kentucky, Lexington, Kentucky
  - William Beaumont Hospital-Troy, Troy, Michigan
  - New York Cardiovascular Associates, New York, New York
  - Unc Hospitals, Department Of Medicine, Chapel Hill, North Carolina
  - Dumc, Durham, North Carolina
  - Carolina Heart Specialists, Gastonia, North Carolina
  - Piedmont Cardiology Associates, Hickory, North Carolina
  - Wake Forest Univ Health Sciences, Winston-Salem, North Carolina
  - Midwest Cardiology Research Foundation, Columbus, Ohio
  - The Dayton Heart Center, Dayton, Ohio
  - Oklahoma Cardiovascular Research Group, Oklahoma City, Oklahoma
  - Geisinger Clinic - Cardiology, Danville, Pennsylvania
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Cardiovascular Associates, P.C, Kingsport, Tennessee
  - University Of Texas Medical School - San Antonio, San Antonio, Texas
  - Tyler Cardiovascular Consultants, Tyler, Texas
  - Virginia Commonwealth University, Richmond, Virginia
- Austria (2):
  - Local Institution, Feldkirch
  - Local Institution, Vienna
- Belgium (7):
  - Local Institution, Huy, Luik
  - Local Institution, Aalst
  - Local Institution, Antwerp
  - Local Institution, Brasschaat
  - Local Institution, Bruges
  - Local Institution, Brussels
  - Local Institution, Genk
- Canada (11):
  - Local Institution, Edmonton, Alberta
  - Local Institution, Victoria, British Columbia
  - Local Institution, St. John's, Newfoundland and Labrador
  - Local Institution, Belleville, Ontario
  - Local Institution, Chatham, Ontario
  - Local Institution, Hamilton, Ontario
  - Local Institution, London, Ontario
  - Local Institution, Oshawa, Ontario
  - Local Institution, Montreal, Quebec
  - Local Institution, Saint-Charles-Borromée, Quebec
  - Local Institution, Terrebonne, Quebec
- Denmark (8):
  - Local Institution, Arhus C
  - Local Institution, Copenhagen
  - Local Institution, Esbjerg
  - Local Institution, Frederiksberg
  - Local Institution, Glostrup Municipality
  - Local Institution, Hellerup
  - Local Institution, Herning
  - Local Institution, Randers
- France (8):
  - Local Institution, Amiens
  - Local Institution, Cholet
  - Local Institution, Dijon
  - Local Institution, Nantes
  - Local Institution, Paris
  - Local Institution, Pessac
  - Local Institution, Roubaix
  - Local Institution, Toulouse
- Germany (8):
  - Local Institution, Berlin
  - Local Institution, Düren
  - Local Institution, Halle
  - Local Institution, Hanover
  - Local Institution, Krefeld
  - Local Institution, Langen
  - Local Institution, Ludwigshafen
  - Local Institution, Witten
- Israel (10):
  - Local Institution, Afula
  - Local Institution, Hadera
  - Local Institution, Haifa
  - Local Institution, Jerusalem
  - Local Institution, Kfar Saba
  - Local Institution, Nazareth
  - Local Institution, Petah Tikva
  - Local Institution, Rehovot
  - Local Institution, Safed
  - Local Institution, Tel Aviv
- Local Institution, Roma, Italy
- Poland (10):
  - Local Institution, Bialystok
  - Local Institution, Bydgoszcz
  - Local Institution, Gdansk
  - Local Institution, Katowice
  - Local Institution, Krakow
  - Local Institution, Lodz
  - Local Institution, Opole
  - Local Institution, Torun
  - Local Institution, Warsaw
  - Local Institution, Zielona Góra
- Russia (6):
  - Local Institution, Kemerovo
  - Local Institution, Moscow
  - Local Institution, Saint Petersburg
  - Local Institution, Saratov
  - Local Institution, Yaroslavl
  - Local Institution, Yaroslav
- Spain (12):
  - Local Institution, Baracaldo (Vizcaya)
  - Local Institution, Barcelona
  - Local Institution, Hospitalet Llobregat Barcelona
  - Local Institution, León
  - Local Institution, Madrid
  - Local Institution, Málaga
  - Local Institution, Oviedo
  - Local Institution, Santiago de Compostela
  - Local Institution, Seville
  - Local Institution, Tarragona
  - Local Institution, Valladolid
  - Local Institution, Villajoyosa
- Sweden (6):
  - Local Institution, Gothenburg
  - Local Institution, Malmo
  - Local Institution, Örebro
  - Local Institution, Stockholm
  - Local Institution, Sundsvall
  - Local Institution, Uppsala
- United Kingdom (8):
  - Local Institution, Stockport, Cheshire
  - Local Institution, Harrow, Middlesex
  - Local Institution, Edinburgh, Midlothian
  - Local Institution, Portadown, Northern Ireland
  - Local Institution, Sheffield, South Yorkshire
  - Local Institution, York, Yorkshire
  - Local Institution, Croydon
  - Local Institution, Leicester

REFERENCES:
- [Derived] APPRAISE Steering Committee and Investigators; Alexander JH, Becker RC, Bhatt DL, Cools F, Crea F, Dellborg M, Fox KA, Goodman SG, Harrington RA, Huber K, Husted S, Lewis BS, Lopez-Sendon J, Mohan P, Montalescot G, Ruda M, Ruzyllo W, Verheugt F, Wallentin L. Apixaban, an oral, direct, selective factor Xa inhibitor, in combination with antiplatelet therapy after acute coronary syndrome: results of the Apixaban for Prevention of Acute Ischemic and Safety Events (APPRAISE) trial. Circulation. 2009 Jun 9;119(22):2877-85. doi: 10.1161/CIRCULATIONAHA.108.832139. Epub 2009 May 26. PMID 19470889

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1741 enrolled; 1715 randomized. Non-randomization reasons: 6 withdrew consent, 1 death, 1 poor/non-compliance, 18 no longer met study criteria. Phase A: placebo and 2 low doses of apixaban; Phase B: placebo, 2 low doses and 2 high doses of apixaban. High dose arms terminated, Phase B continued to enroll participants into placebo and low dose arms.
Groups:
- Placebo: Study was conducted in 2 Phases (A and B). A tablet of Placebo along with ≤ 165 mg of aspirin was given daily for 26 weeks. 75 mg of clopidogrel once a day (QD) was allowed at the investigator's discretion. After 547 subjects were randomized to Phase A, an independent Data and Safety Monitoring Board (DSMB) recommended expanding the randomization to 2 higher doses of apixaban (10 mg BID and 20 mg QD) in Phase B of the study. Approximately 6 months after the start of Phase B, the DSMB recommended apixaban high dose groups be terminated due to excess bleeding in those participants receiving aspirin and clopidogrel concomitantly with high dose apixaban. Treatment and any new randomization into these 2 groups was halted, while randomization and treatment in the placebo and lower dose apixaban groups continued. Follow-up Period started after Week 26 through 30 days after discontinuation of study drug (for treated participants).
- Apixaban 2.5mg BID: In both Phase A and Phase B of the study: Tablet of Apixaban 2.5mg BID for 26 weeks. Also, ≤ 165 mg of aspirin daily. 75 mg of clopidogrel QD was allowed at the investigator's discretion. Follow-up Period started after Week 26 through 30 days after discontinuation of study drug (for treated participants).
- Apixaban 10mg QD: In both Phase A and Phase B of the study: Tablet of Apixaban 10mg QD for 26 weeks. Also, ≤ 165 mg of aspirin daily. 75 mg of clopidogrel QD was allowed at the investigator's discretion. Follow-up Period started after Week 26 through 30 days after discontinuation of study drug (for treated participants).
- Apixaban 10mg BID: Phase B of the Study: Tablet of Apixaban 10mg BID for 26 weeks. Also, ≤ 165 mg of aspirin daily. 75 mg of clopidogrel QD was allowed at the investigator's discretion.
  Approximately 6 months after the start of Phase B, the DSMB recommended that the 10 mg BID QD group, be terminated due to excess bleeding for participants receiving aspirin and clopidogrel concomitantly with the 10 mg BID apixaban. Follow-up Period started after Week 26 through 30 days after discontinuation of study drug (for treated participants).
- Apixaban 20 mg QD: Phase B of the Study: Tablet of Apixaban 20 mg QD for 26 weeks. Also, ≤ 165 mg of aspirin daily. 75 mg of clopidogrel QD was allowed at the investigator's discretion.
  Approximately 6 months after the start of Phase B, the DSMB recommended that the apixaban 20 mg QD group, be terminated due to excess bleeding for participants receiving aspirin and clopidogrel concomitantly with the apixaban. Follow-up Period started after Week 26 through 30 days after discontinuation of study drug (for treated participants).
Period: Randomized in Phase A (26 Weeks)
Arm/Group | Placebo | Apixaban 2.5mg BID | Apixaban 10mg QD | Apixaban 10mg BID | Apixaban 20 mg QD
Started | 184 | 179 | 184 | 0 | 0
Completed | 130 | 140 | 149 | 0 | 0
Not Completed | 54 | 39 | 35 | 0 | 0
Not completed — Adverse Event | 19 | 14 | 17 | 0 | 0
Not completed — Withdrawal by Subject | 20 | 12 | 13 | 0 | 0
Not completed — Death | 3 | 4 | 0 | 0 | 0
Not completed — Lost to Follow-up | 4 | 4 | 2 | 0 | 0
Not completed — Poor/non-compliance | 3 | 2 | 1 | 0 | 0
Not completed — no longer meets criteria | 4 | 3 | 2 | 0 | 0
Not completed — Administrative reason (arm terminated) | 1 | 0 | 0 | 0 | 0
Period: Randomized in Phase B (26 Weeks)
Arm/Group | Placebo | Apixaban 2.5mg BID | Apixaban 10mg QD | Apixaban 10mg BID | Apixaban 20 mg QD
Started | 427 | 138 | 134 | 248 | 221
Start of Phase B to High Dose Terminated | 368 | 120 | 110 | 248 | 221
Completed | 333 | 105 | 94 | 15 | 13
Not Completed | 94 | 33 | 40 | 233 | 208
Not completed — Adverse Event | 34 | 9 | 12 | 23 | 19
Not completed — Withdrawal by Subject | 35 | 14 | 19 | 15 | 19
Not completed — Death | 5 | 3 | 1 | 0 | 1
Not completed — Lost to Follow-up | 5 | 2 | 3 | 2 | 3
Not completed — poor/non-compliance | 3 | 1 | 3 | 0 | 0
Not completed — no longer meets criteria | 9 | 3 | 2 | 0 | 2
Not completed — Administrative reason by Sponsor | 2 | 1 | 0 | 193 | 164
Not completed — non-specified | 1 | 0 | 0 | 0 | 0
Period: Follow-Up(30days)-Randomized Phase A
Arm/Group | Placebo | Apixaban 2.5mg BID | Apixaban 10mg QD | Apixaban 10mg BID | Apixaban 20 mg QD
Started | 163 | 162 | 174 | 0 | 0
Completed | 158 | 156 | 172 | 0 | 0
Not Completed | 5 | 6 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 5 | 5 | 2 | 0 | 0
Not completed — Death | 0 | 1 | 0 | 0 | 0
Period: Follow-Up(30days)-Randomized Phase B
Arm/Group | Placebo | Apixaban 2.5mg BID | Apixaban 10mg QD | Apixaban 10mg BID | Apixaban 20 mg QD
Started | 383 | 123 | 119 | 222 | 201
Completed | 380 | 123 | 117 | 217 | 199
Not Completed | 3 | 0 | 2 | 5 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 2 | 1 | 1
Not completed — Death | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 2 | 1
Not completed — missing end of study status | 1 | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants were summarized.
Groups:
- Placebo: Tablet of Placebo for 26 weeks. Also, ≤ 165 mg of aspirin daily. 75 mg of clopidogrel QD was allowed at the investigator's discretion.
- Apixaban 2.5mg BID: Tablet of Apixaban 2.5mg BID for 26 weeks. Also, ≤ 165 mg of aspirin daily. 75 mg of clopidogrel QD was allowed at the investigator's discretion.
- Apixaban 10mg QD: Tablet of Apixaban 10mg QD for 26 weeks. Also, ≤ 165 mg of aspirin daily. 75 mg of clopidogrel QD was allowed at the investigator's discretion.
- Apixaban 10mg BID: Tablet of Apixaban 10mg BID for 26 weeks. Also, ≤ 165 mg of aspirin daily. 75 mg of clopidogrel QD was allowed at the investigator's discretion.
  Approximately 6 months after the start of Phase B, this treatment group was terminated
- Apixaban 20 mg QD: Tablet of apixaban, oral, for 26 weeks. Also, ≤ 165 mg of aspirin daily. 75 mg of clopidogrel QD was allowed at the investigator's discretion.
  Approximately 6 months after the start of Phase B, this treatment group was terminated.
- Total: Total of all reporting groups
Arm/Group | Placebo | Apixaban 2.5mg BID | Apixaban 10mg QD | Apixaban 10mg BID | Apixaban 20 mg QD | Total
Number analyzed (Participants) | 611 | 317 | 318 | 248 | 221 | 1715
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.5 (11.25) | 61.1 (11.64) | 60.7 (11.35) | 60.3 (11.00) | 60.9 (11.95) | 60.7 (11.38)
Age, Customized [Number; unit: participants]
  Less than (<) 65 years | 374 | 187 | 197 | 165 | 132 | 1055
  Greater than, equal to 65 and < 75 years | 170 | 85 | 82 | 53 | 57 | 447
  Greater than (>) 75 years | 67 | 45 | 39 | 30 | 32 | 213
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 157 | 75 | 86 | 45 | 50 | 413
  Male | 454 | 242 | 232 | 203 | 171 | 1302
Region of Enrollment [Number; unit: participants]
  Russian Federation | 156 | 93 | 82 | 59 | 52 | 442
  United States | 69 | 40 | 44 | 24 | 14 | 191
  United Kingdom | 15 | 7 | 9 | 5 | 5 | 41
  Spain | 36 | 11 | 16 | 17 | 19 | 99
  Canada | 81 | 47 | 44 | 26 | 21 | 219
  Austria | 4 | 2 | 2 | 4 | 2 | 14
  Sweden | 42 | 21 | 24 | 12 | 12 | 111
  Belgium | 20 | 11 | 9 | 10 | 12 | 62
  Poland | 61 | 21 | 19 | 34 | 31 | 166
  Denmark | 16 | 14 | 15 | 5 | 4 | 54
  Israel | 55 | 29 | 32 | 26 | 21 | 163
  France | 21 | 9 | 8 | 8 | 10 | 56
  Germany | 34 | 12 | 14 | 17 | 18 | 95
  Italy | 1 | 0 | 0 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Event Rate of Composite of Adjudicated Major Bleeding and Clinically Relevant Non-Major Bleeding During the Treatment Period- Treated Participants With Placebo or Apixaban Low Doses
Description: Bleeding was assessed using the International Society on Thrombosis and Hemostasis (ISTH) guidelines. Events were adjudicated by the Clinical Events Committee (CEC). Event rate was number of participants with events divided by the number of participants treated, measured as a percentage (%). The primary outcome is based on data for the placebo and 2 apixaban low-dose groups (2.5 mg BID and 10 mg QD) combined across Phase A and Phase B. The analyses of Phase B data across all doses of apixaban are secondary because of the premature termination of the apixaban high-dose groups (10mg BID, 20mg QD) and the resulting lower duration of exposure for these groups.
Time Frame: From first dose of study drug (Day 1) to last dose plus 2 days, up to Year 2 of the Study
Population: Participants who received at least one dose of placebo or low dose apixaban. Due to the premature termination of the 2 apixaban high-dose groups (10 mg BID and 20 mg QD) in Phase B, the primary analyses reported are based on data for the placebo and 2 apixaban low-dose groups (2.5 mg BID and 10 mg QD) combined across Phase A and Phase B.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Placebo: Tablet of Placebo daily for 26 weeks. Also, less than, equal to (≤) 165 mg of aspirin daily. 75 mg of clopidogrel QD was allowed at the investigator's discretion.
Arm/Group | Placebo | Apixaban 2.5mg BID | Apixaban 10mg QD
Number analyzed (Participants) | 599 | 315 | 315
percentage of participants | 3.0 [1.8 to 4.7] | 5.7 [3.4 to 8.9] | 7.9 [5.2 to 11.5]
Statistical Analysis 1: Comparison: Placebo vs Apixaban 2.5mg BID; Test type: Superiority or Other; Adjusted rate difference = 2.2, 95% CI 2-sided [-1.0 to 5.4] — adjusted difference of event rates takes into consideration stratification factors
Statistical Analysis 2: Comparison: Placebo vs Apixaban 10mg QD; Test type: Superiority or Other; Adjusted Rate Difference = 3.8, 95% CI 2-sided [0.4 to 7.3] — adjusted difference of event rates takes into consideration stratification factors

2. Secondary Outcome: Number of Participants With a Composite of Adjudicated Cardiovascular Death, Non-Fatal Myocardial Infarction, Severe Recurrent Ischemia and Non-Hemorrhagic Stroke During the Intended Treatment Period - Randomized Participants
Description: Events were adjudicated by the Clinical Events Committee (CEC). Intended Treatment Period refers to the period starting on the day of randomization and ending 182 days after the day of randomization (for a total period duration of 183 days). Data in this outcome are combined across Phase A and Phase B.
Time Frame: Randomization to 182 days after randomization (183 days)
Population: Participants who randomized to placebo or low dose apixaban are summarized. Due to the premature termination of the 2 apixaban high-dose groups (10 mg BID and 20 mg QD) in Phase B, the analyses reported are based on data for the placebo and 2 apixaban low-dose groups (2.5 mg BID and 10 mg QD) combined across Phase A and Phase B.
Measure: Number; unit: participants
Arm/Group | Placebo | Apixaban 2.5mg BID | Apixaban 10mg QD
Number analyzed (Participants) | 611 | 317 | 318
participants | 53 | 24 | 19
Statistical Analysis 1: Comparison: Placebo vs Apixaban 2.5mg BID; Test type: Superiority or Other; Hazard Ratio (HR) = 0.73, 95% CI 2-sided [0.44 to 1.19]
Statistical Analysis 2: Comparison: Placebo vs Apixaban 10mg QD; Test type: Superiority or Other; Hazard Ratio (HR) = 0.61, 95% CI 2-sided [0.35 to 1.04]

3. Secondary Outcome: Event Rate for Adjudicated All Bleeding Events During the Treatment Period - Treated Participants With Placebo or Apixaban Low Doses
Description: Bleeding was assessed using the International Society on Thrombosis and Hemostasis (ISTH) guidelines. Events were adjudicated by the Clinical Events Committee (CEC). Event rate was number of participants with events divided by the number of participants treated (%). All bleeding events includes major bleeding, clinically relevant non-major bleeding and minor bleeding. Treatment Period refers to the period from first dose through 2 days, or through 30 days for Serious Adverse Event (SAE) tabulations, after discontinuation of study drug. Data in this outcome are combined across Phase A and Phase B.
Time Frame: first dose (Day 1) to last dose plus 2 days (or for SAEs, plus 30 days), up to Year 2 of the Study
Population: Participants who received at least one dose of placebo or low dose apixaban are summarized. The analyses reported are based on data for the placebo and 2 apixaban low-dose groups (2.5 mg BID and 10 mg QD) combined across Phase A and Phase B.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Placebo: Tablet of Placebo daily for 26 weeks. Also, ≤165 mg of aspirin daily. 75 mg of clopidogrel QD was allowed at the investigator's discretion.
Arm/Group | Placebo | Apixaban 2.5mg BID | Apixaban 10mg QD
Number analyzed (Participants) | 599 | 315 | 315
percentage of participants | 10.5 [8.2 to 13.3] | 20.6 [16.3 to 25.5] | 22.5 [18.0 to 27.6]
Statistical Analysis 1: Comparison: Placebo vs Apixaban 2.5mg BID; Test type: Superiority or Other; Adjusted rate difference = 6.6, 95% CI 2-sided [1.8 to 11.3] — adjusted difference of event rates takes into consideration stratification factors
Statistical Analysis 2: Comparison: Placebo vs Apixaban 10mg QD; Test type: Superiority or Other; Adjusted Rate Difference = 10.0, 95% CI 2-sided [4.8 to 15.2] — adjusted difference of event rates takes into consideration stratification factors

4. Secondary Outcome: Number of Participants With a Composite of Adjudicated All-Cause Death, Non-Fatal Myocardial Infarction, Severe Recurrent Ischemia, and Non-Hemorrhagic Stroke During the Intended Treatment Period - Randomized Participants
Description: Events were adjudicated by the Clinical Events Committee (CEC). Event rate was number of participants with events divided by the number of participants treated (%). Intended Treatment Period refers to the period starting on the day of randomization and ending 182 days after the day of randomization (for a total period duration of 183 days). Data in this outcome are combined across Phase A and Phase B
Time Frame: Day of randomization to 182 days after day of randomization (183 days)
Population: Randomized participants were summarized.
Measure: Number; unit: participants
Arm/Group | Placebo | Apixaban 2.5mg BID | Apixaban 10mg QD
Number analyzed (Participants) | 611 | 317 | 318
participants | 54 | 24 | 20
Statistical Analysis 1: Comparison: Placebo vs Apixaban 2.5mg BID; Test type: Superiority or Other; Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.44 to 1.17]
Statistical Analysis 2: Comparison: Placebo vs Apixaban 10mg QD; Test type: Superiority or Other; Hazard Ratio (HR) = 0.63, 95% CI 2-sided [0.37 to 1.07]

5. Secondary Outcome: Event Rate of Confirmed Adjudicated Major Bleeding During the Treatment Period- Treated Participants With Placebo or Apixaban Low Doses
Description: Bleeding was assessed using the ISTH guidelines. Events were adjudicated by the Clinical Events Committee. Event rate was number of participants with events divided by the number of participants treated, measured as a percentage (%).
Time Frame: from first dose (Day 1) to last dose plus 2 days, up to Year 2 of the Study
Population: Participants who received at least one dose of placebo or low dose apixaban were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Apixaban 2.5mg BID | Apixaban 10mg QD
Number analyzed (Participants) | 599 | 315 | 315
percentage of participants | 0.8 [0.3 to 1.9] | 1.6 [0.5 to 3.7] | 1.9 [0.7 to 4.1]
Statistical Analysis 1: Comparison: Placebo vs Apixaban 2.5mg BID; Test type: Superiority or Other; Adjusted rate difference = 0.3, 95% CI 2-sided [-1.3 to 2.0] — adjusted difference of event rates takes into consideration stratification factors
Statistical Analysis 2: Comparison: Placebo vs Apixaban 10mg QD; Test type: Superiority or Other; Adjusted Rate Difference = 0.8, 95% CI 2-sided [-1.1 to 2.7] — adjusted difference of event rates takes into consideration stratification factors

6. Secondary Outcome: Number of Participants With Composite of Adjudicated All-Cause Death, Non-Fatal Myocardial Infarction, Severe Recurrent Ischemia, Non-Hemorrhagic Stroke During the Phase B Adjusted Intended Treatment Period - Participants Randomized in Phase B
Description: Phase B Adjusted Intended Treatment Period=day of randomization and ends on termination date of high dose apixaban, 1-Oct-2007. The analyses of Phase B data across all doses of apixaban are secondary due to the premature termination of the apixaban high dose groups and the lower duration of exposure.
Time Frame: Day of randomization and ends on high dose termination date, 1-Oct-2007
Population: Participants who were concomitantly randomized in Phase B only were summarized (start of Phase B, March 2007, to termination of high doses in Phase B, October 2007) .
Measure: Number; unit: participants
Groups:
- Apixaban 10mg BID: Tablet of Apixaban 10mg BID for 26 weeks. Also, ≤ 165 mg of aspirin daily. 75 mg of clopidogrel QD was allowed at the investigator's discretion.
  Approximately 6 months after the start of Phase B this treatment group was terminated.
- Apixaban 20 mg QD: Tablet of apixaban QD for 26 weeks. Also, ≤ 165 mg of aspirin daily. 75 mg of clopidogrel QD was allowed at the investigator's discretion.
  Approximately 6 months after the start of Phase B this treatment group was terminated.
Arm/Group | Placebo | Apixaban 2.5mg BID | Apixaban 10mg QD | Apixaban 10mg BID | Apixaban 20 mg QD
Number analyzed (Participants) | 368 | 120 | 110 | 248 | 221
participants | 16 | 6 | 4 | 8 | 7
Statistical Analysis 1: Comparison: Placebo vs Apixaban 2.5mg BID; Test type: Superiority or Other; Hazard Ratio (HR) = 1.13, 95% CI 2-sided [0.44 to 2.88]
Statistical Analysis 2: Comparison: Placebo vs Apixaban 10mg QD; Test type: Superiority or Other; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.29 to 2.57]
Statistical Analysis 3: Comparison: Placebo vs Apixaban 10mg BID; Test type: Superiority or Other; Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.30 to 1.66]
Statistical Analysis 4: Comparison: Placebo vs Apixaban 20 mg QD; Test type: Superiority or Other; Hazard Ratio (HR) = 0.72, 95% CI 2-sided [0.30 to 1.74]

7. Secondary Outcome: Event Rate of Composite of Adjudicated Major Bleeding and Clinically Relevant Non-Major Bleeding During the Phase B Adjusted Treatment Period- Treated Participants Randomized in Phase B
Description: Bleeding was assessed using ISTH guidelines. Events were adjudicated by the CEC. Event rate was number of participants with events divided by the number of participants treated, measured as a percentage (%). The analyses of Phase B data across all doses of apixaban are secondary because of the premature termination of the apixaban high-dose groups and the lower duration of exposure. Phase B Adjusted Treatment Period=safety events occurring in the period from first dose through 2 days (or through 30 days for SAE tabulations) after the earliest of last dose date or 1-Oct-2007 (termination date for the 10 mg BID group).
Time Frame: From first dose (Day 1) to last dose, plus 2 days (plus 30 days for SAEs), up to high dose termination, 1 October 2007
Population: Participants randomized in Phase B only who received at least one dose of placebo or apixaban were summarized.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Placebo: Tablet of Placebo, oral, for 26 weeks. Also ≤ 165 mg of aspirin daily. 75 mg of clopidogrel QD was allowed at the investigator's discretion.
Arm/Group | Placebo | Apixaban 2.5mg BID | Apixaban 10mg QD | Apixaban 10mg BID | Apixaban 20 mg QD
Number analyzed (Participants) | 362 | 119 | 108 | 244 | 218
percentage of participants | 0.8 [0.2 to 2.4] | 5.0 [1.9 to 10.7] | 5.6 [2.1 to 11.7] | 7.8 [4.8 to 11.9] | 7.3 [4.3 to 11.6]
Statistical Analysis 1: Comparison: Placebo vs Apixaban 2.5mg BID; Test type: Superiority or Other; Adjusted Rate Difference = 4.0, 95% CI 2-sided [0.0 to 8.1]
Statistical Analysis 2: Comparison: Placebo vs Apixaban 10mg QD; Test type: Superiority or Other; Adjusted Rate Difference = 4.7, 95% CI 2-sided [0.0 to 9.3]
Statistical Analysis 3: Comparison: Placebo vs Apixaban 10mg BID; Test type: Superiority or Other; Adjusted Rate Difference = 7.0, 95% CI 2-sided [3.4 to 10.5]
Statistical Analysis 4: Comparison: Placebo vs Apixaban 20 mg QD; Test type: Superiority or Other; Adjusted Rate Difference = 4.7, 95% CI 2-sided [1.4 to 8.0]

8. Secondary Outcome: Event Rate for Adjudicated All Bleeding Events During the Phase B Adjusted Treatment Period - Treated Participants Randomized in Phase B
Description: Bleeding was assessed using the ISTH guidelines. Events were adjudicated by the CEC. Event rate was number of participants with events divided by the number of participants treated (%). All bleeding events included major bleeding, clinically relevant non-major bleeding and minor bleeding. Phase B Adjusted Treatment Period=safety events occurring in the period from first dose through 2 days (or through 30 days for SAE tabulations) after the earliest of last dose date or 1-Oct-2007 (termination date for the 10 mg BID group).
Time Frame: From first dose (Day 1) to last dose, plus 2 days (plus 30 days for SAEs), up to high dose termination, 1 October 2007
Population: Participants concomitantly randomized in Phase B who received at least one dose of placebo or apixaban were summarized.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Placebo: Tablet of Placebo daily for 26 weeks. Also ≤ 165 mg of aspirin daily. 75 mg of clopidogrel QD was allowed at the investigator's discretion.
Arm/Group | Placebo | Apixaban 2.5mg BID | Apixaban 10mg QD | Apixaban 10mg BID | Apixaban 20 mg QD
Number analyzed (Participants) | 362 | 119 | 108 | 244 | 218
percentage of participants | 6.1 [3.8 to 9.1] | 15.1 [9.2 to 22.8] | 17.6 [10.9 to 26.1] | 24.2 [18.9 to 30.1] | 23.9 [18.4 to 30.1]
Statistical Analysis 1: Comparison: Placebo vs Apixaban 2.5mg BID; Test type: Superiority or Other; Adjusted Rate Difference = 8.3, 95% CI 2-sided [1.8 to 14.9]
Statistical Analysis 2: Comparison: Placebo vs Apixaban 10mg QD; Test type: Superiority or Other; Adjusted Rate Difference = 10.9, 95% CI 2-sided [3.4 to 18.4]
Statistical Analysis 3: Comparison: Placebo vs Apixaban 10mg BID; Test type: Superiority or Other; Adjusted Rate Difference = 17.4, 95% CI 2-sided [11.6 to 23.2]
Statistical Analysis 4: Comparison: Placebo vs Apixaban 20 mg QD; Test type: Superiority or Other; Adjusted Rate Difference = 10.4, 95% CI 2-sided [5.6 to 15.1]

9. Secondary Outcome: Number of Participants With Composite of Adjudicated Cardiovascular Death, Non-Fatal Myocardial Infarction, Severe Recurrent Ischemia, Non-Hemorrhagic Stroke During the Phase B Adjusted Intended Treatment Period - Participants Randomized in Phase B
Description: Phase B Adjusted Intended Treatment Period=day of randomization and ends on 1-Oct-2007. The analyses of Phase B data across all doses of apixaban are secondary due to the premature termination of the apixaban high dose groups and the lower duration of exposure.
Time Frame: Day of randomization up to high dose termination, 1-Oct-2007
Population: Participants who were concomitantly randomized in Phase B were summarized.
Measure: Number; unit: participants
Arm/Group | Placebo | Apixaban 2.5mg BID | Apixaban 10mg QD | Apixaban 10mg BID | Apixaban 20 mg QD
Number analyzed (Participants) | 368 | 120 | 110 | 248 | 221
participants | 16 | 6 | 4 | 8 | 7
Statistical Analysis 1: Comparison: Placebo vs Apixaban 2.5mg BID; Test type: Superiority or Other; Cox Proportional Hazard = 1.13, 95% CI 2-sided [0.44 to 2.88]
Statistical Analysis 2: Comparison: Placebo vs Apixaban 10mg QD; Test type: Superiority or Other; Cox Proportional Hazard = 0.86, 95% CI 2-sided [0.29 to 2.57]
Statistical Analysis 3: Comparison: Placebo vs Apixaban 10mg BID; Test type: Superiority or Other; Cox Proportional Hazard = 0.71, 95% CI 2-sided [0.30 to 1.66]
Statistical Analysis 4: Comparison: Placebo vs Apixaban 20 mg QD; Test type: Superiority or Other; Cox Proportional Hazard = 0.72, 95% CI 2-sided [0.30 to 1.74]

10. Secondary Outcome: Event Rate of Confirmed Adjudicated Major Bleeding During the Phase B Adjusted Treatment Period - Treated Participants Randomized in Phase B
Description: Bleeding was assessed using the ISTH guidelines. Events were adjudicated by the CEC. Event rate was number of participants with events divided by the number of participants treated (%).
Time Frame: From first dose (Day 1) to last dose, plus 2 days (plus 30 days for SAEs), up to high dose termination, 1 October 2007
Population: Participants concomitantly randomized in Phase B who received at least one dose of placebo or apixaban were summarized.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Apixaban 2.5mg BID | Apixaban 10mg QD | Apixaban 10mg BID | Apixaban 20 mg QD
Number analyzed (Participants) | 362 | 119 | 108 | 244 | 218
percentage of participants | 0.0 [0.0 to 1.0] | 0.8 [0.0 to 4.6] | 0.0 [0.0 to 3.4] | 2.9 [1.2 to 5.8] | 4.1 [1.9 to 7.7]
Statistical Analysis 1: Comparison: Placebo vs Apixaban 2.5mg BID; Test type: Superiority or Other; Adjusted Rate Difference = 0.8, 95% CI 2-sided [-0.9 to 2.6]
Statistical Analysis 2: Comparison: Placebo vs Apixaban 10mg BID; Test type: Superiority or Other; Adjusted Rate Difference = 2.9, 95% CI 2-sided [0.6 to 5.1]
Statistical Analysis 3: Comparison: Placebo vs Apixaban 20 mg QD; Test type: Superiority or Other; Adjusted Rate Difference = 4.1, 95% CI 2-sided [1.3 to 6.9]

ADVERSE EVENTS:
Time Frame: Day 1 up to 30 days post last dose of study drug, up to approximately 2 years: A+B treatment groups. March 2007 up to 30 days post last dose in October 2007 (termination of high doses), are presented in Phase B Treatment groups.
Description: Participants treated with at least 1 dose of study drug are presented. Note: during Phase B, high dose apixaban arms (10 mg BID and 20 mg QD) were terminated but participants could continue to be randomized to Placebo, 2.5 mg BID and 10 mg QD apixaban and treated post termination of the high dose arms (October 2007), up to approximately 2 years.
Groups:
- Phase A+B Apixaban 10mg QD: Total Phase A and Phase B participants combined who received at least 1 dose of 10 mg QD apixaban during the study.
- Phase A+B Apixaban 2.5mg BID: Total Phase A and Phase B participants combined who received at least 1 dose of 2.5 mg BID apixaban during the study.
- Phase A+B Placebo: Total Phase A and Phase B participants combined who received at least 1 dose of placebo during the study.
- Phase B Apixaban 10mg BID: Participants treated with at least one dose of 10 mg BID apixaban during Phase B as measured from the start of randomization in Phase B and up to termination of high dose apixaban (October 2007)
- Phase B Apixaban 10mg QD: Participants treated with at least one dose of 10 mg QD apixaban during Phase B as measured from the start of randomization in Phase B and up to termination of high dose apixaban (October 2007)
- Phase B Apixaban 20mg QD: Participants treated with at least one dose of 20 mg QD apixaban during Phase B as measured from the start of randomization in Phase B and up to termination of high dose apixaban (October 2007)
- Phase B Apixaban 2.5mg BID: Participants treated with at least one dose of 2.5 mg BID apixaban during Phase B as measured from the start of randomization in Phase B and up to termination of high dose apixaban (October 2007)
- Phase B Placebo: Participants treated with at least one dose of Placebo during Phase B as measured from the start of randomization in Phase B and up to termination of high dose apixaban (October 2007)
Arm/Group | Phase A+B Apixaban 10mg QD | Phase A+B Apixaban 2.5mg BID | Phase A+B Placebo | Phase B Apixaban 10mg BID | Phase B Apixaban 10mg QD | Phase B Apixaban 20mg QD | Phase B Apixaban 2.5mg BID | Phase B Placebo
Serious Adverse Events (participants affected / at risk) | 72/315 | 73/315 | 125/599 | 55/244 | 22/108 | 36/218 | 19/119 | 56/362
Other Adverse Events (participants affected / at risk) | 122/315 | 101/315 | 175/599 | 84/244 | 30/108 | 67/218 | 22/119 | 80/362
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase A+B Apixaban 10mg QD (N=315) | Phase A+B Apixaban 2.5mg BID (N=315) | Phase A+B Placebo (N=599) | Phase B Apixaban 10mg BID (N=244) | Phase B Apixaban 10mg QD (N=108) | Phase B Apixaban 20mg QD (N=218) | Phase B Apixaban 2.5mg BID (N=119) | Phase B Placebo (N=362)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Arterial restenosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1 | 2 | 1 | 0 | 0 | 1 | 1
Coronary artery restenosis (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Electrocardiogram change (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
In-stent arterial restenosis (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 2 | 0 | 1 | 1 | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 6 | 8 | 11 | 5 | 1 | 3 | 2 | 4
Angina unstable (Cardiac disorders) | 5 | 6 | 14 | 5 | 2 | 3 | 0 | 6
Bladder cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 3 | 0 | 4 | 1 | 0 | 0 | 0 | 3
Cardiac failure chronic (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 1
Eye haemorrhage (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Lichen planus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Peripheral vascular disorder (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wound abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arteriosclerosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Calculus ureteric (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 7 | 6 | 13 | 7 | 2 | 6 | 1 | 8
Coronary artery dissection (Cardiac disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dyskinesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Impaired healing (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Reflux oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 4 | 4 | 3 | 0 | 1 | 1 | 2
Aneurysm (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arteriogram coronary (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Cardiac enzymes increased (Investigations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypomania (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ischaemia (Vascular disorders) | 8 | 4 | 12 | 4 | 2 | 6 | 1 | 5
Myocardial infarction (Cardiac disorders) | 11 | 8 | 24 | 3 | 3 | 1 | 1 | 12
Myocardial ischaemia (Cardiac disorders) | 0 | 1 | 5 | 0 | 0 | 0 | 0 | 4
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pericarditis (Cardiac disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acute prerenal failure (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Barrett's oesophagus (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bundle branch block right (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Campylobacter gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Chest discomfort (General disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Coronary artery occlusion (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dementia Alzheimer's type (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 0
Endocarditis (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myocardial rupture (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 3 | 1 | 0 | 1 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sudden death (General disorders) | 0 | 3 | 4 | 0 | 0 | 0 | 1 | 0
Syncope vasovagal (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tachyarrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Thrombosis (Vascular disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Uterine polyp (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Volvulus (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal symptom (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Angiopathy (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cardiac failure acute (Cardiac disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Colonic polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Death (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Diabetic gastroparesis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1 | 3 | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Haemorrhage (Vascular disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Septic shock (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sudden cardiac death (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Venous thrombosis limb (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 1 | 2 | 1 | 0 | 0 | 0 | 0
Cardiogenic shock (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Catheter site haemorrhage (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Diplopia (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 6 | 2 | 4 | 5 | 3 | 1 | 0 | 2
Peritonsillar abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sick sinus syndrome (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 4 | 3 | 3 | 0 | 1 | 0 | 1 | 2
Atrial flutter (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 3 | 4 | 2 | 0 | 1 | 0 | 1
Cardiac myxoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear haemorrhage (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 2 | 3 | 2 | 0 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Intermittent claudication (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lung injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vascular pseudoaneurysm (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase A+B Apixaban 10mg QD (N=315) | Phase A+B Apixaban 2.5mg BID (N=315) | Phase A+B Placebo (N=599) | Phase B Apixaban 10mg BID (N=244) | Phase B Apixaban 10mg QD (N=108) | Phase B Apixaban 20mg QD (N=218) | Phase B Apixaban 2.5mg BID (N=119) | Phase B Placebo (N=362)
Dizziness (Nervous system disorders) | 18 | 15 | 35 | 10 | 4 | 9 | 3 | 16
Angina pectoris (Cardiac disorders) | 19 | 18 | 31 | 10 | 5 | 11 | 3 | 12
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 24 | 18 | 18 | 16 | 5 | 25 | 4 | 2
Chest pain (General disorders) | 27 | 21 | 52 | 19 | 9 | 14 | 4 | 24
Gingival bleeding (Gastrointestinal disorders) | 11 | 10 | 9 | 15 | 2 | 8 | 4 | 4
Contusion (Injury, poisoning and procedural complications) | 26 | 20 | 20 | 12 | 4 | 10 | 4 | 10
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 16 | 13 | 20 | 3 | 6 | 4 | 4 | 10
Haematoma (Vascular disorders) | 16 | 11 | 10 | 9 | 5 | 9 | 4 | 5
Headache (Nervous system disorders) | 25 | 17 | 30 | 15 | 2 | 6 | 0 | 12
Fatigue (General disorders) | 8 | 13 | 26 | 16 | 1 | 6 | 4 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.